CLINICAL TRIAL: NCT04625933
Title: The Effect of Body Mass Index (BMI) on Inpatient Stroke Rehabilitation Outcome: A Prospective Study From an East-Asian Cohort
Status: Completed | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Jong Sze Chin, Registrar, Tan Tock Seng Hospital
Other Study IDs: NHG-DSRB 2018/01084
Record Dates: First submitted 2020-10-30; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Weight Change, Body; Stroke
Keywords: Body Mass Index; Stroke Rehabilitation
MeSH Terms: conditions — Body Weight Changes; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Research has shown that rehabilitation at almost any Body Mass Index (BMI) level leads to positive functional outcomes. Some data demonstrating that gains are often more rapid at BMI above "normal". The aim of this study is to investigate the association between BMI and the functional progress of all patients admitted to Tan Tock Seng Tertiary Rehabilitation Center.

ELIGIBILITY:
Inclusion Criteria:

* clinical strokes (ischaemic or haemorrhagic) diagnosed by acute neurologists or neurosurgeons and confirmed on computerized tomography (CT) or Magnetic resonance imaging (MRI) brain imaging
* aged 18 years and above
* admitted directly from acute stroke units
* able to provide informed consent by self or by next of kin in incompetence patient
* must receive physical therapy (either physiotherapy, occupational therapy or speech therapy) at least 5 times a week with each session at least 30 minutes

Exclusion Criteria:

* rehabilitation was not the primary reason for the inpatient admission
* failure to complete the rehabilitation program due to either an acute transfer off rehabilitation or a discharge against medical advice
* incomplete or missing Body Mass Index (BMI) or Functional Independence Measure (FIM) data
* patients who were not of Asian ethnicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient admitted to Tan Tock Seng Tertiary Rehabilitation Centre and fulfilled the inclusion criteria within the study period will be consented to the study.
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) on Admission | Functional Independence Measure (FIM) was measured within 72 hours of admission
  Functional Independence Measure (FIM), the main primary outcome measure during rehabilitation was measured within 72 hours of admission and discharge by rehabilitation therapists all of whom were trained and certified in the use of the FIM. The FIM is an 18-item instrument comprising 13 motor items and 5 cognitive items, with each item graded on a 7-point ordinal scale (1 denotes complete dependence and 7 denotes complete independence), including the ability to perform activities of daily living (ADLs) across 6 areas (self-care, sphincter control, transfers, locomotion, communication, and social cognition). Total admission FIM (Ta-FIM) scores, total discharge FIM (Td-FIM) scores (18 - 126), motor FIM (m-FIM) sub-scores (13 - 91) and cognitive FIM (c-FIM) sub-scores (5 - 35), were tabulated.
Functional Independence Measure (FIM) on Discharge | Functional Independence Measure (FIM) was measured within 72 hours of discharge.
  Functional Independence Measure (FIM), the main primary outcome measure during rehabilitation was measured within 72 hours of admission and discharge by rehabilitation therapists all of whom were trained and certified in the use of the FIM. The FIM is an 18-item instrument comprising 13 motor items and 5 cognitive items, with each item graded on a 7-point ordinal scale (1 denotes complete dependence and 7 denotes complete independence), including the ability to perform activities of daily living (ADLs) across 6 areas (self-care, sphincter control, transfers, locomotion, communication, and social cognition). Total admission FIM (Ta-FIM) scores, total discharge FIM (Td-FIM) scores (18 - 126), motor FIM (m-FIM) sub-scores (13 - 91) and cognitive FIM (c-FIM) sub-scores (5 - 35), were tabulated.

SECONDARY OUTCOMES:
Mean Functional Independence Measure (FIM) Gain | Within 72 hours
  Mean FIM gain, calculated as [Td-FIM - Ta-FIM] points
Mean Functional Independence Measure (FIM) efficiency | Through study completion, an average of 1 year
  Mean FIM efficiency, calculated as [FIM gain]/ [rehabilitation length of stay (days)]
Mean Functional Independence Measure (FIM) effectiveness | Within 72 hours
  Mean FIM effectiveness was calculated as FIM gain/(126 points-FIM admission scores) with a value of 0-1.
Body Mass Index (BMI) | Within 72 hours
  All patients had their weight (in kilograms) and height (in meters) measured on admission and discharge by rehabilitation nurses 72 hours after rehabilitation admission and prior to planned rehabilitation discharge. Weight was measured via sitting weighing scales or platform weighing scale for bedbound patients while height was measured with height measuring scale or measured in a supine position with legs outstretched and feet in dorsiflexion at end of bed for bedbound patients. BMI is then calculated as weight /height in meters squared.

CONTACTS AND LOCATIONS:
Overall Officials: SZE CHIN JONG, MD, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No